CLINICAL TRIAL: NCT05781932
Title: Effects of Barbed Suture Continuous Tension Reduction Suture in Dermal Combined With Epidermal Glue on the Healing of Endoscopic Stuck Hole and Scar Formation
Brief Title: Innovative Suture Technique for Endoscopic Hernia Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yizhuo Lu, MD (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Lu, MD, Director, Head of General surgery, Principal Investigator, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-261
Record Dates: First submitted 2023-03-09; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Suture Techniques; Medical Glue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Histoacryl medical tissue glue (Experimental): specification:0.5 ml/piece, main components: n-butyl 2-cyanoacrylate (embutate), pigment (1-hydroxy-4[(toluene)amino]-9,10-anthraquinone), and stabilizers (p-diphenol, sulfur dioxide, phosphoric acid)
  Interventions: Procedure: Dermal barb suture combined with medical glue

INTERVENTIONS:
Procedure: Dermal barb suture combined with medical glue — In the experimental group, after tension reduction and suture were completed, the wound and surrounding skin were wiped clean with normal saline and clean gauze, and the blood accumulated in the wound was squeezed out. Histoacryl medical tissue glue (specification:0.5 ml/piece, main components: n-butyl 2-cyanoacrylate (embutate), pigment (1-hydroxy-4[(toluene)amino]-9,10-anthraquinone), and stabilizers (p-diphenol, sulfur dioxide, phosphoric acid)) were evenly spread on the surgical incision and kept in the butt state for 4 to 6 seconds. After it got solidify and dry, a sterile gauze covered the surgical incision. There was no need to disinfect and change the dressings after the operation. Patients can shower normally on the day after the operation by just avoiding rubbing the incision covered with glue. Patients can move normally 1-2 days after the operation, and the glue film falls off on its own within 5-10 days.

SUMMARY:
The minimally invasive surgical technique represented by endoscopy is one of the most important inventions in the medical field of the 20th century. Laparoscopic surgery is a technique in which a rod-shaped camera and special surgical instruments are inserted into the body cavity (abdominal cavity, chest cavity, etc.) to complete the surgical operation by poking 3-4 holes (0.5-2 cm in size) in the body wall[2]. These holes are known as poke holes, and the closure of poke holes is a technique that every young surgeon must master. Currently, the proportion of endoscopic minimally invasive surgeries, including inguinal hernia repair, has increased widely in China. Currently, most of inguinal hernia repairs at our center are performed laparoscopically. Shortening the suture time and healing time of the stuck hole, improving the healing strength of the skin, and reducing scar hyperplasia are issues worth discussing.

Barbed sutures were first used in plastic surgery and are now widely used in laparoscopic tissue suturing. Because it is knot-free and one-way tightening, the tension of the incision can be released evenly, avoiding excessive local tension in the incision and causing ischemia and necrosis, which in turn affects the healing of the incision. Barbed thread sutures can be used to quickly close the incision and achieve excellent results. A good incision reduces tension and prevents scarring. Medical glue can quickly form a thin waterproof film on the surface of an incision, which promotes blood coagulation, wound shrinkage, and sealing.

Inguinal hernia is a common and frequently occurring condition. Minimally invasive surgery for an inguinal hernia can reduce postoperative pain, help patients resume daily activities early, and achieve rapid recovery; therefore, it is being accepted by an increasing number of people[12]. After laparoscopy, the treatment of poking holes is an indispensable part of surgery and is directly related to postoperative recovery, aesthetics, and patient satisfaction. Combining the continuous tension reduction suture of the dermis barbed suture with epidermis glue should help achieve better incision healing, reduce incision scars, and simultaneously return to daily activities faster, shower after surgery, and improve the medical treatment experience. This is the first study to try this novel approach.

A total of 100 patients who underwent laparoscopic total extraperitoneal (TEP) inguinal hernia repair in the General Surgery Department of Zhongshan Hospital Affiliated with Xiamen University from January 2022 to May 2022 were selected as the research subjects. They were randomly divided into two groups; the traditional Vicryl interrupted suture was used to poke the hole (control group), and the dermis barbed suture was used for continuous tension reduction suture combined with the epidermis glue to poke the hole (experimental group). Statistical differences were compared between the two stitching methods regarding operation time, incision healing, incision healing scars, and incision complications.

ELIGIBILITY:
Inclusion Criteria:

* (1) outpatients diagnosed with inguinal hernia by color Doppler ultrasound or CT examination and
* (2) signed informed consent.

Exclusion Criteria:

* (1) other serious diseases of the system, such as severe cardiopulmonary dysfunction and liver and kidney insufficiency;
* (2) obvious abnormal coagulation function;
* (3) history of open lower abdominal surgery;
* (4) inability to complete follow-up or treatment compliance;
* (5) high risk of incision infection.

Ages: 46 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
During surgery | The time required to close the abdominal wall incision
  The time of suturing the punch hole was recorded.
Surgical incision healing | 2 weeks after the operation,
  the wound healing grading standard (grade A healing: the incision healed well without adverse reactions; grade B healing: inflammation, such as redness and swelling at the wound healing site. , induration but not suppuration; Grade C healing: incision suppuration, incision, and drainage are required).
Scar scoring | Three months after the operation,
  Vancouver scar scale (VSS).The VSS mainly evaluates the color, thickness, softness, and vascular distribution of scars, with a total score of 15 points, with higher scores indicating more severe scars.
Pain score: | 1 week after the operation
  According to the corresponding numbers, pain can be divided into different degrees: grade 0, no pain, grade 1-3, mild pain; grade 4- Grade 6 is moderate pain; and grades 7-10, severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Yizhuo Lu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No